CLINICAL TRIAL: NCT05846321
Title: Registry for Vascular Trauma and Follow-up Examinations
Status: Recruiting | Type: Observational
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Other Study IDs: Vascular Registry
Record Dates: First submitted 2023-03-15; First posted 2023-05-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-03

CONDITIONS: Vascular Injury
Keywords: Trauma; Vascular trauma; Bleeding; Ischemia; Registry
MeSH Terms: conditions — Vascular System Injuries; Wounds and Injuries; Hemorrhage; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Within the framework of the project presented here, a registry for traumatic vascular injuries will be established at Augsburg University Hospital. Patients who are treated at our hospital for an isolated vascular trauma or a vascular involvement in (poly-)trauma will be included. This is a rare complication of trauma, so data collection in a registry is useful to pool data on therapeutic procedures and outcome.

These patients differ from the usual vascular surgery patient clientele because there is usually no previous vascular disease. Healthy vessels show different physiological responses than pre-diseased vessels. The usual therapeutic procedures and materials are also developed for arteriosclerotic or aneurysmatic vessels. Therefore, a core objective of this study is to assess long-term outcomes after vascular trauma.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Vascular involvement in trauma
* Isolated vascular injury
* Written informed consent, except for those deceased from trauma sequelae

Exclusion Criteria:

* Minority
* Lack of consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated at university hospital Augsburg for trauma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Long term follow-up after vascular injury | Assessments will be performed at different time points. In the first year after trauma at 3 time points: 3, 6 and 12 months. Through study completion, an average of 1 year
  Inclusion of patients in the vascular trauma registry, then regular follow-up examinations.
  Conditions resulting from the trauma are to be assessed and recorded. Therefore several examinations should be performed.
  The kind of examination is due to trauma localization an treatment.
  Most examinations are non invasive as ultrasound, ABI-measurement and clinical evaluation.
  Ultrasound documents the patency of vessels/grafts (primary outcome measure). ABI-measurement ist documented as Index (primary outcome measure) Some patients require CT- or MRI-Scans for example in the follow-up of aortic stentgrafts, they document graft patency, vessel diameter in centimeters and endoleak formation (primary outcome measure).
  The abovementioned examinations combined document the graft/vessel patency as primary outcome measure

SECONDARY OUTCOMES:
Reintervention rate | Assessments will be performed at different time points. In the first year after trauma at 3 time points: 3, 6 and 12 months. Through study completion, an average of 1 year
  Treatment of complications as graft occlusion or stenosis
Development of treatment patterns | Assessments will be performed at different time points. In the first year after trauma at 3 time points: 3, 6 and 12 months. Through study completion, an average of 1 year
  Optional, depending on the amount and quality of data

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Augsburg, Augsburg, Germany